CLINICAL TRIAL: NCT02989194
Title: A Phase 2a Double-blind, Placebo-controlled Study to Assess the Safety and Tolerability of a Single Intravenous Dose of an Investigational Monoclonal Antibody With Code Name VIS410 in Subjects With Uncomplicated Influenza A Infection
Brief Title: Study of an Investigational Monoclonal Antibody, VIS410, in Subjects With Uncomplicated Influenza A
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Visterra, Inc. (Industry)
Collaborators: Biomedical Advanced Research and Development Authority (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIS410-202
Record Dates: First submitted 2016-12-05; First posted 2016-12-12 (Estimated); Results first posted 2022-08-15 (Actual); Last update posted 2022-08-15 (Actual); Status verified 2022-08

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- VIS410 low dose (Experimental): Single intravenous fixed low dose of VIS410
  Interventions: Drug: VIS410 low dose
- VIS410 high dose (Experimental): Single intravenous fixed high dose of VIS410
  Interventions: Drug: VIS410 high dose
- Placebo (Placebo Comparator): Single intravenous placebo infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VIS410 low dose — Single intravenous fixed low dose of VIS410
  Arms: VIS410 low dose
Drug: VIS410 high dose — Single intravenous fixed high dose of VIS410
  Arms: VIS410 high dose
Drug: Placebo — Single intravenous infusion of placebo
  Arms: Placebo

SUMMARY:
This is a Phase 2a randomized, double-blind, placebo-controlled study designed to assess the safety and tolerability of an investigational monoclonal antibody, VIS410, in subjects with uncomplicated influenza.

DETAILED DESCRIPTION:
Subjects will be admitted to an infusion unit for drug administration and observation following infusion. The study is designed to compare an infusion of a single high or low IV dose of VIS410 against placebo. Subjects will be followed for 100 (±7 days).

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged ≥18 years and ˂65 years
* Women should fulfill one of the following criteria:

  1. Post-menopausal; either amenorrhea ≥12 months or follicle stimulating hormone >40 mIU/mL (milli-international units/milliliter) as documented in their medical history
  2. Surgically sterile; hysterectomy, bilateral oophorectomy, or tubal ligation
  3. Women of childbearing potential participating in heterosexual sexual relations must be willing to use adequate contraception from screening until 60 days post infusion
* Non-vasectomized (or vasectomized less than 6 months prior to dosing) male subjects who have a female partner of childbearing potential must use an effective birth control method when having heterosexual intercourse, from screening until 60 days post infusion
* Test positive for influenza A by Rapid Antigen Test performed with a commercially available test on an adequate nasopharyngeal specimen in accordance with the manufacturer's instructions
* Presence of at least one respiratory symptom (cough, sore throat, or nasal symptoms) of moderate to severe intensity, or presence of at least one constitutional symptom (myalgia [aches and pains], headache, feverishness, or fatigue) of moderate to severe intensity
* Onset of symptoms (time when the temperature was first measured as elevated [temperature of ≥100.4°F or ≥38°C], OR the time when the subject experienced at least one respiratory symptom or at least one constitutional symptom) no more than 72 hours before the start of infusion

Exclusion Criteria:

* Use of NSAIDs or antihistamines within 6 hours of study drug dosing with the exception of those used as part of the pretreatment regimen
* History of intolerance or allergic response to monoclonal antibodies and/or pretreatment medications (diphenhydramine, ibuprofen and acetylsalicylic acid)
* Subject weight less than (<) 45 kg
* Subjects with clinical history that would lead to increased risk of influenza complications including but not limited to clinically significant cardiac disease, moderate to severe asthma, or other moderate to severe chronic obstructive pulmonary disease, metabolic syndrome including moderate to severe diabetes or active tuberculosis
* History of chronic GI disease, including bleeding, ulceration, Irritable Bowel Syndrome, systemic mastocytosis or chronic diarrhea
* Women who are pregnant, breast-feeding, or considering becoming pregnant
* Patients with hypoxemia requiring oxygen support
* Clinical evidence of worsening of any chronic medical condition (temporally associated with the onset of symptoms of influenza) which, in the Investigator's opinion, indicates that such finding(s) could represent complications of influenza
* Presence of immunocompromised status due to chronic illness, previous organ transplant, or use of immunosuppressive medical therapy including systemic steroids
* Presence of known Acquired Immune Deficiency Syndrome-defining illness, chronic hepatitis B or hepatitis C
* Receipt of any dose of antiviral therapy such as, but not limited to, rimantadine, amantadine, peramivir, zanamivir, laninamivir or oseltamivir in the 7 days prior to screening
* Enrollment in any other investigational drug or device study, any disease or vaccine study within 30 days prior to Day 1 or within 5 half-lives of the investigational compound, whichever is longer
* Subjects unable to take oral predose medication
* Known or suspected alcohol or drug abuse, that is, abuse of a level that would compromise the safety or cooperation of the subject in the opinion of the Investigator
* Subjects on chronic medications where the dose has not been stable for at least 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2017-10-27 (Actual); Study Completion 2017-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Visterra, Inc.
Locations (46):
- United States (10):
  - Huntsville, Alabama
  - Coral Gables, Florida
  - Homestead, Florida
  - Miami, Florida
  - Orlando, Florida
  - Eunice, Louisiana
  - New Orleans, Louisiana
  - Shelby, North Carolina
  - Houston, Texas
  - McAllen, Texas
- Bulgaria (5):
  - Asenovgrad
  - Lom
  - Rousse
  - Sofia
  - Velingrad
- Estonia (2):
  - Paide
  - Tallinn
- Latvia (6):
  - Daugavpils
  - Liepāja
  - Rēzekne
  - Riga
  - Valmiera
  - Ventspils
- Serbia (3):
  - Kragujevac
  - Niš
  - Novi Sad
- South Africa (15):
  - Welkom, Free State
  - Benoni, Gauteng
  - Centurion, Gauteng
  - Johannesburg, Gauteng
  - Kempton Park, Gauteng
  - Pretoria, Gauteng
  - Pretoria West, Gauteng
  - Soshanguve, Gauteng
  - Soweto, Gauteng
  - Durban, KwaZulu-Natal
  - Thabazimbi, Limpopo
  - Middelburg, Mpumalanga
  - Witbank, Mpumalanga
  - Cape Town, Western Cape
  - Worcester, Western Cape
- Ukraine (5):
  - Kharkiv
  - Kiev
  - Odesa
  - Sumy
  - Vinnytsia

IPD SHARING:
Plan to Share IPD: No
No plans to share IPD

REFERENCES:
- [Result] Hershberger E, Sloan S, Narayan K, Hay CA, Smith P, Engler F, Jeeninga R, Smits S, Trevejo J, Shriver Z, Oldach D. Safety and efficacy of monoclonal antibody VIS410 in adults with uncomplicated influenza A infection: Results from a randomized, double-blind, phase-2, placebo-controlled study. EBioMedicine. 2019 Feb;40:574-582. doi: 10.1016/j.ebiom.2018.12.051. Epub 2019 Jan 9. PMID 30638863

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was initiated in 58 study centers; 28 sites enrolled at least 1 subject.
Pre-assignment Details: When required, subject may have been given a pre-screening informed consent to perform a Rapid Antigen Test for influenza. Flu-positive subjects were given a full explanation of the nature of the study and written informed consent (approved by local ethics committee) was obtained according to local requirements before any study related assessments
Groups:
- VIS410 High Dose: Single intravenous fixed dose of 4000 mg VIS410
- VIS410 Low Dose: Single intravenous fixed dose of 2000 mg VIS410
- Placebo: Single intravenous saline solution
Period: Overall Study
Arm/Group | VIS410 High Dose | VIS410 Low Dose | Placebo
Started | 50 | 50 | 50
Completed | 49 | 48 | 50
Not Completed | 1 | 2 | 0
Not completed — Study on hold for safety and participant was withdrawn | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VIS410 High Dose | VIS410 Low Dose | Placebo | Total
Number analyzed (Participants) | 50 | 50 | 50 | 150
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 50 | 150
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (13.13) | 39.6 (13.79) | 43.1 (12.77) | 41.0 (13.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 29 | 28 | 84
  Male | 23 | 21 | 22 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 12 | 13 | 35
  Not Hispanic or Latino | 40 | 38 | 37 | 115
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 11 | 10 | 31
  White | 38 | 38 | 36 | 112
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 3 | 4
Region of Enrollment [Number; unit: participants]
  Latvia | 6 | 2 | 7 | 15
  United States | 19 | 21 | 18 | 58
  South Africa | 24 | 25 | 24 | 73
  Estonia | 1 | 2 | 0 | 3
  Bulgaria | 0 | 0 | 1 | 1
Subjects Body Mass Index [Mean (Full Range); unit: kg/m^2] | 29.01 [19.4 to 48.0] | 30.80 [16.7 to 55.6] | 28.82 [18.0 to 43.1] | 29.54 [16.7 to 55.6]
Time since onset of influenza (hours) [Mean (Standard Deviation); unit: hours] — Population: Participant was omitted if the date/time of symptom onset was missing.
  hours
    number analyzed (Participants) | 49 | 49 | 50 | 148
    (all) | 43.31 (16.479) | 40.57 (11.563) | 38.19 (13.859) | 40.67 (14.170)
Time since onset of influenza (hours) [Median (Full Range); unit: hours] — Median time since onset of influenza in hours. Population: Participants who did not have a start date/time for symptom onset were excluded.
  hours
    number analyzed (Participants) | 49 | 49 | 50 | 148
    (all) | 27.69 [19.4 to 48.0] | 28.88 [16.7 to 55.6] | 28.07 [18.0 to 43.1] | 28.60 [16.7 to 55.6]

OUTCOME MEASURES:

1. Primary Outcome: Assess the Safety and Tolerability of a Single IV Dose of VIS410 in Participants With Uncomplicated Influenza Infection
Description: The percentage of participants with adverse events (AEs) and serious adverse events (SAEs) following administration of a single dose of IV VIS410.
Time Frame: 100 days
Population: Safety Population The safety population included all subjects randomized who received IV study drug. The safety population summaries were based on the actual treatment received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- VIS410 High Dose: Single intravenous dose of 4000 mg VIS410
- VIS410 Low Dose: Single intravenous dose of 2000 mg VIS410
- VIS410 Total: Summation of the VIS410 high and low dose groups.
- Placebo: Single intravenous dose of saline solution
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 49 | 49 | 98 | 50
percentage of participants
  Percentage of subjects with any adverse events | 57.1 [42.21 to 71.18] | 34.7 [21.67 to 49.64] | 45.9 [35.80 to 56.29] | 26.0 [14.63 to 40.34]
  Percentage of subjects with any serious adverse events | 0 [0.00 to 7.25] | 0 [0.00 to 7.25] | 0 [0.0 to 3.69] | 4 [0.49 to 13.71]

2. Primary Outcome: Percentage of Participants With Any Treatment-emergent Adverse Event (TEAE) and TEAEs of Special Interest
Description: Percentage of participants experiencing any TEAE, TEAEs considered related to study treatment and the number of participants experiencing adverse events of special interest (AESI). A TEAE is defined as an adverse event that starts on or after the date of study drug IV infusion. AESIs included hypersensitivity reaction, anaphylactic reaction, or injection site adverse event.
Time Frame: 100 days
Population: Safety Population. The safety population included all participants randomized who received IV study drug. The safety population summaries were based on the actual treatment received.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Total VIS410: Summation of 4000 mg and 2000 mg VIS410 dose groups.
Arm/Group | VIS410 High Dose | VIS410 Low Dose | Total VIS410 | Placebo
Number analyzed (Participants) | 49 | 49 | 98 | 50
percentage of participants
  Percentage of subjects with any TEAE | 55.1 [40.23 to 69.33] | 34.7 [21.67 to 49.64] | 44.9 [34.83 to 55.28] | 24.0 [13.06 to 38.17]
  Percentage of subjects with treatment related TEAEs | 30.6 [18.25 to 45.42] | 14.3 [5.94 to 27.24] | 22.4 [14.64 to 31.99] | 12.0 [4.53 to 24.31]
  Percentage of subjects with any TEAEs of Special Interest | 34.7 [21.67 to 49.64] | 16.3 [7.32 to 29.66] | 25.5 [17.24 to 35.31] | 12 [4.53 to 24.31]
  Percentage of Subjects with any hypersensitivity Reactions | 0 [0.00 to 7.25] | 0 [0.00 to 7.25] | 0 [0.00 to 3.69] | 0 [0.00 to 7.11]
  Percentage of subjects with any anaphylactic reactions | 0 [0.00 to 7.25] | 0 [0.00 to 7.25] | 0 [0.00 to 3.69] | 0 [0.00 to 7.11]
  Percentage of subjects with any injection site AEs. | 2.0 [0.05 to 10.85] | 0.0 [0.00 to 7.25] | 1.0 [0.03 to 5.55] | 0 [0.00 to 7.11]

3. Secondary Outcome: Percentage Change From Baseline in Signs and Symptoms of Influenza-like Illness as Assessed by the Influenza Patient Reported Outcomes Questionnaire After a Single IV Dose of VIS410
Description: The Influenza Patient Reported Outcome (FluPRO) questionnaire is a 32-question instrument that assesses the occurrence and intensity of influenza associated symptoms (scale of 0 to 4, with 0 representing no symptoms) over 24 hours (lower scores indicate better outcomes). FluPRO data were recorded by subjects at Baseline (Day 1), then daily thereafter through Day 10. These data were summarized at each visit by treatment group. The data below show the percent change in mean total symptom scores over time by treatment arm.
Time Frame: 10 days
Population: Modified Intent-to-Treat Population. The modified intent-to-treat (mITT) population included all subjects who received IV study drug and were confirmed influenza A positive by a molecular test at the central virological laboratory.
Measure: Mean (Standard Deviation); unit: Percent Change
Groups:
- VIS410 Total: Summation of the 4000 and 2000 mg dose groups
- Placebo: Single dose intravenous saline solution
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 46 | 44 | 90 | 48
Percent Change
  Percent Change from Baseline to Day 2 | -26.12 (27.00) | -29.98 (29.55) | -28.01 (28.18) | -19.53 (26.51)
  Percentage change from baseline to day 3 | -38.65 (28.78) | -49.37 (29.62) | -43.89 (29.53) | -33.63 (23.60)
  Percentage change from baseline to day 4 | -53.46 (26.16) | -59.08 (31.12) | -56.21 (28.67) | -44.55 (28.20)
  Percentage change from baseline to day 5 | -60.85 (25.52) | -64.61 (29.91) | -62.69 (27.66) | -56.75 (24.31)
  Percentage change from baseline to day 6 | -69.31 (20.90) | -66.80 (33.42) | -68.08 (27.61) | 64.01 (23.35)
  Percentage change from baseline to day 7 | -74.03 (19.31) | -70.76 (31.18) | -72.43 (25.71) | -71.51 (20.61)
  Percentage change from baseline to day 8 | -77.98 (20.76) | -76.03 (25.53) | -77.02 (23.13) | -76.16 (21.01)
  Percentage change from baseline to day 9 | -80.05 (19.78) | -78.48 (25.95) | -79.27 (22.91) | -79.52 (19.84)
  Percentage change from baseline to day 10 | -82.30 (20.07) | -81.38 (20.43) | -81.85 (20.14) | -84.35 (17.52)
Statistical Analysis 1: Comparison: VIS410 Total vs Placebo; Percent Change from Baseline to Day 2. All null hypotheses were defined as no treatment difference; Test type: Superiority — Descriptive statistics. All statistical comparisons were performed using 2-sided tests at the 0.05 significance level; p = 0.158, Wilcoxon (Mann-Whitney) — All p-values are presented for informational purposes only, there were no adjustments for multiple comparisons
Statistical Analysis 2: Comparison: VIS410 Total vs Placebo; Percent Change from Baseline to Day 3. All null hypotheses were defined as no treatment difference; Test type: Superiority — Descriptive statistics. All statistical comparisons were performed using 2-sided tests at the 0.05 significance level; p = 0.025, Wilcoxon (Mann-Whitney) — All p-values are presented for informational purposes only, there were no adjustments for multiple comparisons
Statistical Analysis 3: Comparison: VIS410 Total vs Placebo; Percent Change from Baseline to Day 4. All null hypotheses were defined as no treatment difference; Test type: Superiority — Descriptive statistics. All statistical comparisons were performed using 2-sided tests at the 0.05 significance level; p = 0.007, Wilcoxon (Mann-Whitney) — All p-values are presented for informational purposes only, there were no adjustments for multiple comparisons
Statistical Analysis 4: Comparison: VIS410 Total vs Placebo; Percent Change from Baseline to Day 5. All null hypotheses were defined as no treatment difference; Test type: Superiority — Descriptive statistics. All statistical comparisons were performed using 2-sided tests at the 0.05 significance level; p = 0.061, Wilcoxon (Mann-Whitney) — All p-values are presented for informational purposes only, there were no adjustments for multiple comparisons
Statistical Analysis 5: Comparison: VIS410 Total vs Placebo; Percent Change from Baseline to Day 6. All null hypotheses were defined as no treatment difference; Test type: Superiority — Descriptive statistics. All statistical comparisons were performed using 2-sided tests at the 0.05 significance level; p = 0.107, Wilcoxon (Mann-Whitney) — All p-values are presented for informational purposes only, there were no adjustments for multiple comparisons
Statistical Analysis 6: Comparison: VIS410 Total vs Placebo; Percent Change from Baseline to Day 7. All null hypotheses were defined as no treatment difference; Test type: Superiority — Descriptive statistics. All statistical comparisons were performed using 2-sided tests at the 0.05 significance level; p = 0.237, Wilcoxon (Mann-Whitney) — All p-values are presented for informational purposes only, there were no adjustments for multiple comparisons
Statistical Analysis 7: Comparison: VIS410 Total vs Placebo; Percent Change from Baseline to Day 8. All null hypotheses were defined as no treatment difference; Test type: Superiority — Descriptive statistics. All statistical comparisons were performed using 2-sided tests at the 0.05 significance level; p = 0.497, Wilcoxon (Mann-Whitney) — All p-values are presented for informational purposes only, there were no adjustments for multiple comparisons
Statistical Analysis 8: Comparison: VIS410 Total vs Placebo; Percent Change from Baseline to Day 9. All null hypotheses were defined as no treatment difference; Test type: Superiority — Descriptive statistics. All statistical comparisons were performed using 2-sided tests at the 0.05 significance level; p = 0.704, Wilcoxon (Mann-Whitney) — All p-values are presented for informational purposes only, there were no adjustments for multiple comparisons
Statistical Analysis 9: Comparison: VIS410 Total vs Placebo; Percent Change from Baseline to Day 10. All null hypotheses were defined as no treatment difference; Test type: Superiority — Descriptive statistics. All statistical comparisons were performed using 2-sided tests at the 0.05 significance level; p = 0.585, Wilcoxon (Mann-Whitney) — All p-values are presented for informational purposes only, there were no adjustments for multiple comparisons

4. Secondary Outcome: Hospitalization for Influenza-related Complications
Description: Number of participants requiring hospitalization for influenza-related complications
Time Frame: 100 days
Population: Modified Intent-to-Treat Population The modified intent-to-treat (mITT) population included all subjects who received IV study drug and were confirmed influenza A positive by a molecular test at the central virological laboratory.
Measure: Count of Participants; unit: Participants
Groups:
- VIS410 Total: Summation of 4000 and 2000 mg VIS410 dose groups
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 46 | 44 | 90 | 48
Participants | 0 | 0 | 0 | 0

5. Secondary Outcome: Duration of Hospitalization for Complications of Influenza
Description: Duration of hospitalization for participants with at least 1 complication of influenza. There were no participants hospitalized for complications of influenza.
Time Frame: 100 days
Population: as for outcome 3
Measure: Number; unit: days
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 46 | 44 | 90 | 48
days | 0 | 0 | 0 | 0

6. Secondary Outcome: Count of Participants With Complications of Influenza
Description: Count of participants with at least 1 complication of influenza
Time Frame: 100 days
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 46 | 44 | 90 | 48
participants | 1 [0.06 to 11.53] | 3 [1.43 to 18.66] | 4 [1.22 to 10.99] | 3 [1.31 to 17.2]

7. Secondary Outcome: Influenza A Relapse/Reinfection
Description: Number of participants with influenza A relapse/reinfection
Time Frame: 100 days
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 46 | 44 | 90 | 48
Participants | 0 | 0 | 0 | 0

8. Secondary Outcome: VIS410 Maximum Plasma Concentration
Description: The maximum observed concentration of VIS410 in serum (Cmax).
Time Frame: 1, 3, 5, 7, 14, 28, 56, 100 days
Population: The Pharmacokinetics (PK) population included all subjects who received IV study drug and had at least 1 PK concentration that could be calculated
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | VIS410 High Dose | VIS410 Low Dose
Number analyzed (Participants) | 47 | 49
mcg/mL | 1013.559 (35.5) | 627.640 (54.6)

9. Secondary Outcome: Pharmacokinetics of VIS410 Concentration in Serum
Description: Time corresponding to the maximum serum concentration of VIS410.
Time Frame: 1, 3, 5, 7, 14, 28, 56, 100 days
Population: The PK population included all subjects who received IV study drug and had at least 1 PK concentration that could be calculated
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day
Arm/Group | VIS410 High Dose | VIS410 Low Dose
Number analyzed (Participants) | 47 | 49
day | 0.119 (79.0624) | 0.133 (131.4255)

10. Secondary Outcome: VIS410 Plasma Concentration ( AUC 0-infinity)
Description: VIS410 area under the plasma concentration time curve in serum. AUC 0-infinity is from the time of dosing extrapolated to infinity.
Time Frame: 1, 3, 5, 7, 14, 28, 56, 100 days
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*mcg/mL
Arm/Group | VIS410 High Dose | VIS410 Low Dose
Number analyzed (Participants) | 46 | 48
day*mcg/mL | 8598.909 (38.3172) | 5371.988 (30.0631)

11. Secondary Outcome: VIS410 Plasma Concentration (AUC 0-last)
Description: VIS410 area under the plasma concentration time curve in serum. AUC 0-last is the area under the plasma concentration time curve from time 0 to the last measurable concentration.
Time Frame: 1, 3, 5, 7, 14, 28, 56, 100 days
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*mcg/mL
Arm/Group | VIS410 High Dose | VIS410 Low Dose
Number analyzed (Participants) | 47 | 49
day*mcg/mL | 8441.244 (39.5852) | 5385.491 (31.2065)

12. Secondary Outcome: Half-life of VIS410 in Serum.
Description: Terminal elimination half-life of VIS410 in serum (t1/2) in serum.
Time Frame: 1, 3, 5, 7, 14, 28, 56, 100 days
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day
Arm/Group | VIS410 High Dose | VIS410 Low Dose
Number analyzed (Participants) | 46 | 48
day | 9.941 (40.6241) | 10.119 (34.2559)

13. Secondary Outcome: Clearance (CL) of VIS410 in Serum.
Description: Summary of VIS410 total clearance (CL) in serum.
Time Frame: 1, 3, 5, 7, 14, 28, 56, 100 days
Population: as for outcome 9
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mL/day
Arm/Group | VIS410 High Dose | VIS410 Low Dose
Number analyzed (Participants) | 46 | 48
mL/day | 465.175 (38.3172) | 372.302 (30.0631)

14. Secondary Outcome: Area Under the Viral Load-Time Curve (VL AUC) From Nasopharyngeal Swab Day 7.
Description: The difference between VIS410 and placebo treatment groups in viral AUC based on the half-maximal tissue culture infective dose (TCID50) from nasopharyngeal swab samples taken from the first 50 participants.
Time Frame: 7 days
Population: as for outcome 4
Measure: Median (Full Range); unit: d x log10 TCID50/mL
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 46 | 44 | 90 | 48
d x log10 TCID50/mL | 3.726 [0.15 to 14.44] | 3.570 [0.14 to 13.37] | 3.660 [0.14 to 14.44] | 4.782 [0.28 to 16.57]
Statistical Analysis 1: Comparison: VIS410 Total vs Placebo; A t-test was used to assess the difference between the VIS410 total and placebo treatment groups from nasopharyngeal swabs based on the TCID50; Test type: Superiority — All statistical comparisons were performed using 2-sided tests at the 0.05 significance level; p = 0.083, t-test, 2 sided

15. Secondary Outcome: Peak Viral Load by TCID50
Description: The difference between VIS410 and placebo treatment groups in peak viral load based on the half-maximal tissue culture infective dose (TCID50) from nasopharyngeal swab samples taken from the first 50 participants.
Time Frame: 7 days
Population: as for outcome 4
Measure: Median (Full Range); unit: log10 TCID50/mL
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 46 | 44 | 90 | 48
log10 TCID50/mL | 3.125 [0.38 to 5.75] | 2.50 [0.38 to 4.75] | 2.625 [0.38 to 5.75] | 3.375 [0.38 to 6.75]
Statistical Analysis 1: Comparison: VIS410 Total vs Placebo; The null hypothesis was defined as no treatment difference; Test type: Superiority — All statistical comparisons were performed using 2-sided tests at the 0.05 significance level; p = 0.169, t-test, 2 sided — All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons

16. Secondary Outcome: Time to Resolution of Peak Viral Load From Nasopharyngeal Samples by TCID50.
Description: The number of days for the median time to resolution of peak viral load from end of infusion by nasopharyngeal swabs collected from the first 50 participants and tested by half maximal tissue culture infective dose (TCID50)
Time Frame: 7 days
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: days
Groups:
- VIS649 Total: Summation of 4000 and 2000 mg VIS410 dose groups.
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS649 Total | Placebo
Number analyzed (Participants) | 46 | 44 | 90 | 48
days | 2.0 [1.81 to 2.90] | 1.9 [1.83 to 2.87] | 1.9 [1.84 to 2.10] | 3.6 [1.83 to 3.85]
Statistical Analysis 1: Comparison: VIS649 Total vs Placebo; Kaplan-Meier methods were used to calculate the median time. All null hypotheses were defined as no treatment difference; Test type: Superiority — Descriptive Statistics. Statistical comparisons were performed using log rank test; p = 0.028, Log Rank — All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons; All statistical comparisons were performed using 2-sided tests at the 0.05 significance level, unless specifically stated otherwise. All null hypotheses were defined as no treatment difference. All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons

17. Secondary Outcome: Summary of Anti-VIS410 Antibody (ADA) Titers.
Description: Count of subjects testing positive for anti-VIS410 antibodies on days 1, 14, 56 and 100. A positive result includes samples confirmed positive and above titer cut point factor (and titer ≥ 1). Negative results include screened or confirmed negative or confirmed positive but below titer cut point factor (titer < 1). For participants receiving placebo, only samples from two participants were tested at Days 14 and 56.
Time Frame: 100 days
Population: Safety Population The safety population included all ITT subjects who received IV study drug. The safety population summaries were based on the actual treatment received. Not all participants had samples for all timepoints. For participants receiving placebo, all participants were tested on Day 1 and Day 100; only samples from two participants were tested at Days 14 and 56.
Measure: Count of Participants; unit: Participants
Groups:
- VIS410 Total: All participants receiving VIS410
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 49 | 49 | 98 | 50
Participants
  Visit day 1 anti-VIS410 antibody titer: number analyzed (Participants) | 49 | 47 | 96 | 49
  Visit day 1 anti-VIS410 antibody titer: ADA Titer ≤ 1 | 45 | 43 | 88 | 45
  Visit day 1 anti-VIS410 antibody titer: ADA Titer > 1 to 4 | 3 | 3 | 6 | 4
  Visit day 1 anti-VIS410 antibody titer: ADA Titer > 4 to 16 | 1 | 1 | 2 | 0
  Visit day 1 anti-VIS410 antibody titer: ADA Titer > 16 to 64 | 0 | 0 | 0 | 0
  Visit day 1 anti-VIS410 antibody titer: ADA Titer > 64 | 0 | 0 | 0 | 0
  Day 14 anti-VIS410 antibody titer: number analyzed (Participants) | 49 | 47 | 96 | 2
  Day 14 anti-VIS410 antibody titer: ADA Titer ≤ 1 | 46 | 43 | 89 | 1
  Day 14 anti-VIS410 antibody titer: ADA Titer > 1 to 4 | 2 | 3 | 5 | 1
  Day 14 anti-VIS410 antibody titer: ADA Titer > 4 to 16 | 1 | 1 | 2 | 0
  Day 14 anti-VIS410 antibody titer: ADA Titer > 16 to 64 | 0 | 0 | 0 | 0
  Day 14 anti-VIS410 antibody titer: ADA Titer > 64 | 0 | 0 | 0 | 0
  Day 56 anti-VIS410 antibody titer: number analyzed (Participants) | 49 | 48 | 97 | 2
  Day 56 anti-VIS410 antibody titer: ADA Titer ≤ 1 | 42 | 34 | 76 | 2
  Day 56 anti-VIS410 antibody titer: ADA Titer > 1 to 4 | 5 | 8 | 13 | 0
  Day 56 anti-VIS410 antibody titer: ADA Titer > 4 to 16 | 1 | 3 | 4 | 0
  Day 56 anti-VIS410 antibody titer: ADA Titer > 16 to 64 | 1 | 3 | 4 | 0
  Day 56 anti-VIS410 antibody titer: ADA Titer > 64 | 0 | 0 | 0 | 0
  Day 100 anti-VIS410 antibody titer: number analyzed (Participants) | 49 | 47 | 96 | 50
  Day 100 anti-VIS410 antibody titer: ADA Titer ≤ 1 | 32 | 26 | 58 | 47
  Day 100 anti-VIS410 antibody titer: ADA Titer > 1 to 4 | 6 | 8 | 14 | 3
  Day 100 anti-VIS410 antibody titer: ADA Titer > 4 to 16 | 10 | 11 | 21 | 0
  Day 100 anti-VIS410 antibody titer: ADA Titer > 16 to 64 | 1 | 2 | 3 | 0
  Day 100 anti-VIS410 antibody titer: ADA Titer > 64 | 0 | 0 | 0 | 0

18. Secondary Outcome: Duration of Signs and Symptoms of Influenza-like Illness as Assessed by the Influenza Patient Reported Outcomes Questionnaire After a Single IV Dose of VIS410
Description: The Influenza Patient Reported Outcome (FluPRO) questionnaire is a 32-question instrument that assesses the occurrence and intensity of influenza associated symptoms (scale of 0 to 4, with 0 representing no symptoms) over 24 hours (lower scores indicate better outcomes). FluPRO data were recorded by subjects at Baseline (Day 1), then daily thereafter through Day 10. Data below show the time to symptom resolution for Total Symptom Score.
Time Frame: 10 days
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | VIS410 High Dose | VIS410 Low Dose | VIS410 Total | Placebo
Number analyzed (Participants) | 46 | 44 | 90 | 48
days | 2.7 [1.4 to 4.1] | 2.0 [1.0 to 3.0] | 2.1 [1.0 to 3.8] | 2.6 [1.3 to 4.0]
Statistical Analysis 1: Comparison: VIS410 Total vs Placebo; All null hypotheses were defined as no treatment difference; Test type: Equivalence — Descriptive Statistics. All statistical comparisons were performed at the 0.05 significance level; p = 0.173, Log Rank — All p-values are presented for informational purposes only; there were no adjustments for multiple comparisons; Kaplan-Meier methods were used to calculate the median time, 25th percentile and 75th percentile

ADVERSE EVENTS:
Time Frame: Adverse events were monitored continuously from signing of informed consent until the last study related activity (100 days).
Description: New or worsening symptoms of influenza, including cough, sore throat, nasal congestion, fatigue, headache, myalgia or low-grade fever were in general, considered a component of the presenting illness, and were not reported as AEs unless they resulted in an SAE
Arm/Group | VIS410 High Dose | VIS410 Low Dose | Placebo
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49 | 2/50
Other Adverse Events (participants affected / at risk) | 16/49 | 10/49 | 7/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VIS410 High Dose (N=49) | VIS410 Low Dose (N=49) | Placebo (N=50)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VIS410 High Dose (N=49) | VIS410 Low Dose (N=49) | Placebo (N=50)
Diarrhea (Gastrointestinal disorders) | 13 (13) | 8 (8) | 6 (6)
Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-03-14): https://cdn.clinicaltrials.gov/large-docs/94/NCT02989194/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-05): https://cdn.clinicaltrials.gov/large-docs/94/NCT02989194/SAP_001.pdf